CLINICAL TRIAL: NCT04161937
Title: Work-site Intervention Study to Prevent Diabetes in Nepal
Acronym: WSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Prajjwal Pyakurel, Assistant Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35/2017; BLSCHP-1603 (Other Grant/Funding Number: Bernard Lown Scholar for Cardiovascular Health Program); 5DP1ES02545903 (Other Grant/Funding Number: NIH Director's Pioneer Award)
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Diabetes
Keywords: Work-site; Diabetes; Nepal
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: We have intervention and control arm and at the same time parellel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioural Intervention (Experimental): Half of the randomly selected participants will get behavioural intervention based on Diabetes Prevention Program module.The behavioural intervention classed will be administered by trained nurse weekly for 16 weeks.After completion of behavioural intervention both the experimental and control arm will get cafeteria intervention.
  Interventions: Behavioral: Behavioural Intervention
- Control (Experimental): Half of the participants will act as a control and will not receive any form of behavioural intervention.
  Interventions: Behavioral: Behavioural Intervention

INTERVENTIONS:
Behavioral: Behavioural Intervention — Behavior intervention will comprise of combination of intensive education session, group counseling, goal setting and monitoring based on the Diabetes Prevention Program (DPP).The curriculum includes 24 sessions: 16 core sessions weekly during the first four months of the program followed by a monthly maintenance sessions.

SUMMARY:
The burden of non-communicable disease is on the rise in low- and middle- income countries.Cardiovascular disease is the leading cause of morbidity, mortality, and disability in South Asian regions. Diabetes mellitus is among the top five risk factors for cardiovascular deaths in the world.

Despite the evidence supporting the use of lifestyle interventions to prevent diabetes and improve glucose tolerance, their translation in real world has been challenging. Work-site-based health programs have shown positive impacts on employee health, and have shown significant improvements in blood glucose levels and HbA1C.

The research will be conducted in 1) Hulas wire Industry and 2) Pragati Textile Industry Private limited.

Investigator will conduct before-and-after intervention among pre-diabetic employees.In addition screening will be done to identify the eligible participants.Those who are pregnant,under diabetic and hypertensive medication will be excluded from the study. All of the interested adult employees (≥18 years) will be invited for the first screening. All individuals with HbA1C from 5.7% to 6.4 % will be invited to participate in the study. At baseline, investigators will administer a standardized questionnaire to record the characteristics of the participants.Blood samples will be collected and analyzed for HbA1c, fasting glucose, and lipid profile.

Investigators will have a wait period before implementing any intervention.After completion of control period,half of the participants will be randomized to receive behavioral interventions. Behavior intervention will comprise of combination of intensive education session, group counseling, goal setting and monitoring.Trained nurses will deliver the sessions once every week for two months and then once every month.All the participants will receive canteen intervention after behavioral intervention which will comprise of promotion of healthy foods in the canteen of the study site i.e Improve physical facility ,increase access to healthy food, Information, Education and communication, changes in food price and training of canteen staffs Investigators will conduct follow up at 6 months, 12 months, and 18 months and if funds are available at 24 months. During each follow up, the proportion of unhealthy diet consumption data will be abstracted. In addition, blood samples will be collected and analyzed for HbA1c, fasting glucose, and lipid profile .This period will serve as control group.

DETAILED DESCRIPTION:
Diabetes is the fifth leading cause of death in the most high-income countries and there is substantial evidence that it is epidemic in many low- and middle-income countries. Complications from diabetes, such as coronary artery and peripheral vascular disease, stroke, diabetic neuropathy, amputations, renal failure and blindness results in disability, reduced life expectancy and enormous health costs.The global age standardized prevalence of diabetes has nearly doubled since 1980, rising from 4.7% to 8.5% in the adult population.In Nepal, there is a lack of reliable and representative data on the prevalence of type 2 diabetes.Various small studies from different parts of the country have shown prevalence rates ranging from 6.3% to 8.5%.The burden of diabetes in terms of disability adjusted life years has increased almost 100% from 1990 to 2010. A pilot study in an industrial setting showed a prevalence of 4% diabetes and 31% pre-diabetes among adult employees.The prevention of type 2 diabetes through lifestyle intervention has been established by several clinical trials.These studies had a strong focus on increased physical activity and dietary modification as well as weight reduction among overweight participants. The US Diabetes Prevention Program clinical trial demonstrated that structured lifestyle interventions-such as training people with pre-diabetes to achieve modest weight loss through diet and physical activity-reduced three-year diabetes incidence by 58 percent. Studies have shown that simple modifications to the physical environment can be important in increasing physical activity and altering dietary habits. However, the translation of the knowledge to the real world setting is a challenge. Strategies to translate the preventive measures by innovative and culturally specific environmental and individual level intervention are lacking.

Work-site could be an effective platform to translate this knowledge into action as employed adults spend most of their workday waking hours at workplaces.Workplaces have additional advantages because of convenience to reach people; social support; existing formal and informal communication networks; and possible corporate behavior network.Studies have shown positive impact of diabetes prevention at work-site and other settings.Additionally,environmental changes to the work-sites can achieve modest improvement in employees' health risks, including weight and body mass index ( BMI) measures, in one year and reduced glycated hemoglobin(HbA1c) among pre-diabetic adult employee. In 2013, investigators conducted a survey of cardiovascular disease risk factors among employees of a wire industry in the eastern Nepal. The study showed that about a third of the employees were pre-diabetic and 4% had diabetes. Investigators established an ongoing work-site screening and preventive cardiovascular disease care program in the wire industry in January 2016. Furthermore, investigators conducted a qualitative study to understand willingness, facilitators and barriers to promote healthy diet in the industry cafeteria (unpublished). Building on these ground works, investigators propose implementing and evaluating the effectiveness of a work-site based lifestyle modification - an environmental modification in cafeterias and a lifestyle change education package.Investigators propose a pre-post trial with a control period to assess the effectiveness of the individual level lifestyle intervention on diabetes risk reduction among pre-diabetic (HbA1c of 5.7 to 6.4%) employees of two industries in Nepal.Investigators will provide lifestyle education to half of the randomly selected participants after 6 to 14 months of control period. Additionally, cafeteria intervention will be provided to all the pre-diabetic participants. The study aims to:

Aim 1: To measure the effectiveness of an environmental-level cafeteria intervention on diabetes risk.

Aim 2: To measure the effectiveness of an individual-level lifestyle education on the risk of diabetes prevention.

If the program is shown to be effective at these work-sites, the results of this study will be used to recommend and disseminate a sustainable environment and lifestyle interventions at work-sites to improve the health of workers, other Nepali work-sites, and to Nepal's national program for prevention and control of non- communicable disease. Furthermore, lessons from this study can be used to make recommendations or plan studies of similar work-site programs in the U.S. and other settings outside of Nepal.

ELIGIBILITY:
Inclusion Criteria:

1) Pre-diabetic participants (HbA1c 5.7-6.4%) and FBS (>=100 to 125mg/dl)

Exclusion Criteria:

1. Diabetic - HbA1c (>=6.5%) and FBS > 126mg/dl
2. HbA1c <5.7% and FBS <100mg/dl
3. Taking hypertension,diabetes medication
4. Pregnancy
5. Temporary workers
6. Age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 24months
  The primary outcome is absolute change in HbA1c

CONTACTS AND LOCATIONS:
Locations (1):
- Hulas Wire industry Private Limited and Pragati Textile Industry Private Limited, Biratnagar, Provinve 1, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
We will decide later on

REFERENCES:
- [Derived] Pyakurel P, Shrestha A, Karmacharya BM, Budhathoki SS, Chaudhari RK, Tamrakar D, Shrestha A, Karmacharya RM, Shrestha A, Sharma S, Sharma SK, Spiegelman D. Worksite intervention study to prevent diabetes in Nepal: a randomised trial protocol. Open Heart. 2020 Aug;7(2):e001236. doi: 10.1136/openhrt-2019-001236. PMID 32847993